CLINICAL TRIAL: NCT05262517
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Safety and Efficacy Trial of BHV-3000 (Rimegepant) Orally Disintegrating Tablet (ODT) for the Acute Treatment of Temporomandibular Disorders (TMD)
Brief Title: Safety and Efficacy of BHV-3000 (Rimegepant) Orally Disintegrating Tablet for Acute Treatment of Temporomandibular Disorders
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision to discontinue the study based on adjusted clinical development plan. This decision is not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3000-317; C4951016 (Other: Alias Study Number)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular Disorders; TMD; Temporomandibular Joint; TMJ
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV3000 (rimegepant) (Experimental): One dose of rimegepant 75 mg ODT
  Interventions: Drug: Rimegepant
- Matching Placebo (Placebo Comparator): One dose of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — 75 mg ODT
  Other Names: BHV3000
  Arms: BHV3000 (rimegepant)
Drug: Placebo — matching placebo
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of rimegepant versus placebo in the acute treatment of Temporomandibular Disorders (TMD), which are medical conditions involving the temporomandibular joint (the joint connecting the jawbone to the skull) and surrounding muscles and tissues.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a minimum 3-month to a maximum 5-year history of temporomandibular disorder diagnosed by a healthcare provider.

* At least one instance of pain ≥ 6 on a Numeric Rating Scale (NRS) (0-10) in the jaw and/or temple area on either side in the past 30 days prior to the Screening Visit.
* Subject agrees to study-required restrictions of new pain medication, injection therapy, oral devices, occlusal splint therapy or any other pain management techniques during the course of the study.
* Subject agrees to study-required birth control methods during the course of the study and female subjects must not be breastfeeding.
* No clinically significant abnormality identified on the medical or laboratory evaluation.

Exclusion Criteria:

* Subject has an exclusionary headache, joint, pain, connective tissue, or developmental disorder.

* Subject has an exclusionary history of trauma, surgery, or radiation treatment to the head and neck.
* Body Mass Index ≥ 33kg/m2.
* Subject history of exclusionary medical conditions such as HIV disease, cardiovascular conditions, uncontrolled hypertension or diabetes, psychiatric conditions, drug or alcohol abuse, malignancies, drug allergies, or any significant and/or unstable medical conditions.
* Subjects taking/using excluded therapies.
* Participation in clinical trial with non-biological investigational agents or investigational interventional treatments.
* Subjects who have previously participated in any BHV-3000/ BMS-927711/ rimegepant study.
* Planned participation in any other investigational clinical trial while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (32):
  - Bruce Nelson, DDS, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - The Medici Medical Research, LLC, Hollywood, Florida
  - The Medici Medical Research, Hollywood, Florida
  - SouthCoast Research Center, Inc, Miami, Florida
  - SouthCoast Research Center, Miami, Florida
  - Oceane7 Medical & Research Center, Inc., Miami, Florida
  - Florida Craniofacial Institute, Tampa, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Campus Health, Indiana University-Purdue University Indianapolis, Indianapolis, Indiana
  - IDS-IU Simon Cancer Center (IUSCC), Indianapolis, Indiana
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - University of Kentucky, College of Dentistry, Lexington, Kentucky
  - TMD, Orofacial Pain and Dental Sleep Medicine Clinic, School of Dentistry, University of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Clinvest Research, LLC, Springfield, Missouri
  - Clinvest Research, Springfield, Missouri
  - North Suffolk Neurology, Commack, New York
  - University of Rochester, Rochester, New York
  - Duke University, Raleigh, North Carolina
  - META Medical Research Institute,LLC., Dayton, Ohio
  - Meta Medical Research, Dayton, Ohio
  - Kulkarni Orthodonties, Springboro, Ohio
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Red Star Research, LLC, Lake Jackson, Texas
  - Red Star Research, Lake Jackson, Texas
  - FMC Science, Lampasas, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - JBR, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Snoring and Sleep Apnea Center (DC/TMD Exam - Dr. Christian), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 participants were enrolled in the study. Only 87 participants were randomized to treatment and only 71 participants were treated.
Pre-assignment Details: Participants were to administer one dose of study medication only when temporomandibular disorders (TMD)-associated pain in the jaw and/or temple area on either side reached pain intensity of greater than or equal to (>=) 6 on the numeric rating scale (NRS) in the electronic (e)-diary within 45 days of randomization.
Groups:
- Rimegepant (BHV3000): Participants were randomized for administration of rimegepant 75 milligram (mg) single dose as orally disintegrated tablet (ODT) sublingually.
- Placebo: Participants were randomized for administration of single dose of placebo matching to rimegepant.
Period: Overall Study
Arm/Group | Rimegepant (BHV3000) | Placebo
Started | 44 | 43
Treated | 39 | 32
Completed | 39 | 32
Not Completed | 5 | 11
Not completed — Randomized but not treated | 5 | 11

BASELINE CHARACTERISTICS:
Population: Analysis population included participants who were enrolled and received at least 1 dose of study medication. Baseline characteristics tabulated by the treated analysis set.
Groups:
- Rimegepant (BHV3000): Participants were randomized for administration of rimegepant 75 mg single dose as ODT sublingually.
- Total: Total of all reporting groups
Arm/Group | Rimegepant (BHV3000) | Placebo | Total
Number analyzed (Participants) | 39 | 32 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (13.93) | 38.6 (12.53) | 41.1 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 21 | 49
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 36 | 30 | 66
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) From Baseline to 2-Hours Post-dose (SPID-2)
Description: The SPID-2 was calculated by multiplying the pain intensity difference (PID) score at each post-dose timepoint by the duration (in hours) since the preceding timepoint, then summing the values over the 2 hours. Participants indicated pain using e-diary at each timepoint (0, 15, 30, 45-, 60-, 90- and 120-minutes post-dose) on an NRS score ranging from 0 (no pain) to 10 (worst imaginable pain). PID: calculated by finding the difference between the NRS score at each timepoint from the baseline NRS score (PID range is -6 [best] to 4 [worst]). Assuming a baseline pain intensity score of 6, possible score range of SPID-2 was: -12 (best) to 8 (worst). Lower SPID-2 score = more improvement from pain. SPID-2 Best is 2 hours*-6 = -12 (assuming 0 pain intensity score [pain-free] for each timepoint) and 2) Worst is 2 hours*4 = 8 (assuming 10 pain intensity score [worst imaginable pain] for each timepoint).
Time Frame: Baseline (0 hours) to 2-hours post-dose
Population: Treated analysis population included enrolled participants who took study therapy (rimegepant or placebo); i.e., non-missing study drug start date. Missing postbaseline NRS assessments were imputed as the last non-missing observation prior to the missing assessment. Missing baseline assessments were imputed as the mean of the non-missing baseline assessments across participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Units on a scale | -3.82 [-5.12 to -2.51] | -3.67 [-5.14 to -2.20]
Statistical Analysis 1: Comparison: Rimegepant (BHV3000) vs Placebo; LS means and CIs were estimated by an analysis of covariance (ANCOVA) model, using restricted maximum likelihood (REML) with baseline NRS value as a covariate and treatment group and stratification factor (use of daily medications/ oral devices to reduce the intensity of TMD symptoms) as the main effects; Test type: Other; Least square (LS) mean difference = -0.15, 95% CI 2-sided [-1.78 to 1.48]

2. Primary Outcome: SPID From Baseline to 24-Hours Post-dose (SPID-24)
Description: The SPID-24 was calculated by multiplying the PID score at each post-dose timepoint by the duration (in hours) since the preceding timepoint, then summing the values over the 24 hours. Participants indicated pain using e-diary at each timepoint (0, 15, 30, 45, 60, 90 and 120 minutes and 4-, 8-, and 24-hours post-dose) on an NRS score ranging from 0 (no pain) to 10 (worst imaginable pain). PID: calculated by finding the difference between the NRS score at each timepoint from the baseline NRS score (PID range is -6 [best] to 4 [worst]). Assuming a baseline pain intensity score of 6, possible score range of SPID-24 was: -144 (Best) to 96 (worst). Lower SPID-24 score = more improvement from pain. SPID-24 best and worst scores were calculated as: 1) Best is 24 hours* -6 = -144 (assuming 0 pain intensity score for each timepoint) and 2) Worst is 24 hours*4 = 96 (assuming 10 pain intensity score for each timepoint).
Time Frame: Baseline (0 hours) to 24-hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Unit on a scale | -104.66 [-125.89 to -83.44] | -109.79 [-133.65 to -85.92]
Statistical Analysis 1: Comparison: Rimegepant (BHV3000) vs Placebo; LS means and CIs were estimated by an analysis of covariance model using REML with baseline NRS value as a covariate and treatment group and stratification factor (use of daily medications/ oral devices to reduce the intensity of TMD symptoms) as the main effects; Test type: Other; LS mean difference = 5.12, 95% CI 2-sided [-21.35 to 31.59]

3. Secondary Outcome: Change From Baseline in NRS Score at 2-Hours Post-Dose
Description: TMD pain was assessed using an NRS score ranging in integers from 0 to 10, with 0 being "no pain" and 10 being "worst imaginable pain."
Time Frame: Baseline (0 hours), 2-hours post-dose
Population: Treated analysis population included enrolled participants who took study therapy (rimegepant or placebo); i.e., non-missing study drug start date.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Units on a scale | -3.08 [-3.89 to -2.26] | -3.28 [-4.19 to -2.38]
Statistical Analysis 1: Comparison: Rimegepant (BHV3000) vs Placebo; LS means, and CIs were based on a generalized linear mixed effect model (GLMEM) that included the baseline value as a covariate and fixed effects for treatment group, stratification factor (use of daily medications/ oral devices to reduce the intensity of TMD symptoms; yes or no), scheduled time point, and time point by-treatment group interaction; Test type: Other; LS mean difference = 0.21, 95% CI 2-sided [-0.99 to 1.41]

4. Secondary Outcome: Percentage of Participants Who Experienced Pain Freedom at 2-Hours Post-Dose
Description: Pain freedom was defined as an NRS score of zero at 2 hours post-dose (yes or no). TMD pain was assessed using an NRS score ranging in integers from 0 to 10, with 0 being "no pain" and 10 being "worst imaginable pain."
Time Frame: Baseline (0 hour) to 2-hours post-dose
Population: Treated analysis population included enrolled participants who took study therapy (rimegepant or placebo); i.e., non-missing study drug start date. Participants who (1) had missing data at 2-hours post-dose or (2) took rescue medication at or before 2-hours post-dose were imputed as failures.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Percentage of participants | 10.3 [0.7 to 19.8] | 15.6 [3.0 to 28.2]
Statistical Analysis 1: Comparison: Rimegepant (BHV3000) vs Placebo; Stratified by use of daily medications/ oral devices to reduce the intensity of TMD symptoms at randomization with Mantel-Haenzsel weighting; Test type: Other; Difference in percentage = -5.2, 95% CI 2-sided [-21.3 to 10.9]

5. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Time to onset of meaningful pain relief post-dose is defined as the first nominal timepoint at which a 30% reduction of pain from baseline on NRS is achieved. TMD pain was assessed using an NRS score ranging in integers from 0 to 10, with 0 being "no pain" and 10 being "worst imaginable pain." Kaplan-Meier method was used for analysis.
Time Frame: Baseline (0 hours) up to 24 hours post-dose
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Minutes | 91.3 [56.0 to 233.6] | 120.3 [62.4 to 233.2]

6. Secondary Outcome: Time to Onset of Initial Pain Relief
Description: Time to onset of initial pain relief post-dose is defined as the first nominal timepoint at which a 1-point reduction of pain from baseline on NRS is achieved. TMD pain was assessed using an NRS score ranging in integers from 0 to 10, with 0 being "no pain" and 10 being "worst imaginable pain." Kaplan-Meier method was used for analysis.
Time Frame: Baseline (0 hour) to 24 hours post-dose
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Minutes | 45.3 [30.5 to 54.7] | 45.2 [26.0 to 57.8]

7. Secondary Outcome: Percentage of Participants Using Rescue Medication Within 24 Hours Post-Dose
Description: Rescue medications included any non-study medication recorded on the rescue medication case report form (CRF) with complete medication dates, and either (1) medication date/time is after the study drug start date/time if the medication time and study drug start time are both not missing, or (2) medication date is on or after study drug start date if the medication time or study drug start time is missing.
Time Frame: Through 24 hours post-dose
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant (BHV3000) | Placebo
Number analyzed (Participants) | 39 | 32
Percentage of participants | 10.3 [0.7 to 19.8] | 6.3 [0.0 to 14.6]
Statistical Analysis 1: Comparison: Rimegepant (BHV3000) vs Placebo; Stratified by use of daily medications/oral devices to reduce the intensity of TMD symptoms at randomization with Mantel-Haenszel weighting; Test type: Other; Difference in percentage = 4.0, 95% CI 2-sided [-8.7 to 16.6]

ADVERSE EVENTS:
Time Frame: Randomization up to 7 days after study medication administration (maximum up to 52 days, if study medication took on 45th day post randomization, single dose was to be administered on any day from randomization to 45 days post randomization, only when NRS>=6)
Description: Treated analysis set evaluated.
Arm/Group | Rimegepant (BHV3000) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/32
Other Adverse Events (participants affected / at risk) | 1/39 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant (BHV3000) (N=39) | Placebo (N=32)
Bundle branch block right (Cardiac disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT05262517/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT05262517/SAP_001.pdf